CLINICAL TRIAL: NCT03601195
Title: Prediction of Spontaneous Preterm Birth in Multiple Gestation by Cervical Elastogram
Brief Title: Prediction of Spontaneous Preterm Birth by Cervical Elastogram
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHENG Kwun Yue Yvonne, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CRE 2017.265
Record Dates: First submitted 2018-04-11; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Preterm Birth
Keywords: Sonoelastography
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Chinese women carrying multiple pregnancies

SUMMARY:
Background: Preterm birth is the leading cause of perinatal morbidity and mortality in multiple pregnancies. The medical and educational expenditure and lost productivity associated with preterm birth is very high. Sonoelastography is a new ultrasound technology which has enabled the measurement of tissue stiffness and it has been widely applied in assessment of breast lump and liver cirrhosis. Sonoelastography is potentially useful for the objective assessment of cervical consistency which could be related to risk of preterm birth.

Objective: To assess the cervical consistency by shear wave elastography in prediction of preterm birth in multiple pregnancies.

Setting: This is a prospective non-interventional observational study.

Subjects: Chinese women carrying multiple pregnancies attending antenatal visit are invited to join the study.

Method: Demographic data and antenatal history will be obtained. Transvaginal scan for the cervix will be performed by a trained researcher or obstetrician for the assessment of cervical consistency, cervical length, posterior cervical angle and fetal viability. The measurements will be repeated during 5 antenatal visits or separate study visits at 11-15, 16-19, 20-23, 24-27 and 28-32 weeks of gestation. At the end of pregnancy, the delivery data and neonatal outcome will be collected.

Sample Size: The risk of preterm birth <34 weeks in twin pregnancies is approximately 20%. A sample size of 120 was determined as being sufficient to test the diagnostic performance of cervical elasticity in mid trimester assuming that the risk of preterm delivery <34 weeks vs >34 weeks is 1:5 and that cervical elasticity area under curve (AUC) of the receiver operating characteristics (ROC) curve was 0.7, with 80% power and alpha of 5%.

Data Analysis: Changes in the cervical elastography will be compared using the Student paired two-tailed t test, and in the case of unequal standard deviation (SD), using a Wilcoxon signed-rank paired two-tailed test. For comparison of frequencies, Chi-square test, or a two-sided Fisher exact test will be used where appropriate. Linear regression will be used to assess the correlations. The level of statistical significance is set at p<0.05 (two-sided).

DETAILED DESCRIPTION:
Preterm birth is the leading cause of perinatal morbidity and mortality in multiple pregnancies. The medical and educational expenditure and lost productivity associated with preterm birth is very high. The risk of preterm delivery in singleton pregnancy is 5-7%, and that in twin pregnancy is 7-8 fold higher than singleton pregnancy. Identification of pregnant women at risk of preterm birth could allow intervention to reduce their risk. Sonoelastography is a new ultrasound technology which has enabled the measurement of tissue stiffness and it has been widely applied in assessment of breast lump and liver cirrhosis. Sonoelastography is potentially useful for the objective assessment of cervical consistency which could be related to risk of preterm birth.

Objective:

To assess the cervical consistency by shear wave elastography in prediction of preterm birth in multiple pregnancies.

This is a prospective non-interventional observational study at a university hospital. Chinese women carrying multiple pregnancies attending antenatal visit are invited to participate the study. After informed consent, demographic data and antenatal history of the subjects will be obtained. Transvaginal scan for the cervix will be performed for the assessment of cervical consistency, cervical length, posterior cervical angle and fetal viability. The measurements will be repeated during 5 antenatal visits or separate study visits at 11-15, 16-19, 20-23, 24-27 and 28-32 weeks of gestation. At the end of pregnancy, the delivery data and neonatal outcome will be collected.

Sample Size:

The risk of preterm birth <34 weeks in twin pregnancies is approximately 20%. A sample size of 120 was determined as being sufficient to test the diagnostic performance of cervical elasticity in mid trimester assuming that the risk of preterm delivery <34 weeks vs >34 weeks is 1:5 and that cervical elasticity area under curve (AUC) of the receiver operating characteristics (ROC) curve was 0.7, with 80% power and alpha of 5%.

Data Analysis:

Changes in the cervical elastography will be compared using the Student paired two-tailed t test, and in the case of unequal standard deviation (SD), using a Wilcoxon signed-rank paired two-tailed test. For comparison of frequencies, Chi-square test, or a two-sided Fisher exact test will be used where appropriate. Linear regression will be used to assess the correlations. The level of statistical significance is set at p<0.05 (two-sided).

Implication of data:

A significant improvement in the prediction of preterm delivery allows accurate differentiation of those women who would benefit from treatment for prevention of preterm birth in multiple pregnancies. This would avoid unnecessary intervention, reduce maternal and fetal complications, and has a potential to save medical cost.

ELIGIBILITY:
Inclusion Criteria:

* Chinese women carrying multiple pregnancies attending antenatal visit are invited to join the study.

Exclusion Criteria:

* an age of less than 18 years;
* non-Chinese;
* inability to provide consent;
* refuse to join.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women.
Study Population: Chinese women carrying multiple pregnancies.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-07-02 (Estimated); Study Completion 2019-07-02 (Estimated)

PRIMARY OUTCOMES:
The association of cervical consistency in mid trimester with spontaneous preterm birth in women carrying multiple pregnancies | Between 11 and 32 weeks of gestation
  Cervical consistency will be measured by sonoelastography in term of kilopascals.

SECONDARY OUTCOMES:
The change in cervical consistency during pregnancy in women carrying multiple pregnancies | Between 11 and 32 weeks of gestation
  Cervical consistency will be measured by sonoelastography in term of kilopascals.

CONTACTS AND LOCATIONS:
Overall Officials: Tak Yeung LEUNG, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03601195/Prot_SAP_000.pdf